CLINICAL TRIAL: NCT06324994
Title: A Single-arm, Open-label, National Multi-center Clinical Study of Linperlisib in Combination With Obinutuzumab and Venetoclax in the Treatment of Relapsed and Refractory Blastoid Variant of Mantle Cell Lymphoma (R/R BV-MCL)
Brief Title: Linperlisib Plus Obinutuzumab and Venetoclax for Relapsed and Refractory Blastoid Variant of Mantle Cell Lymphoma.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dalian Medical University (Other)
Responsible Party: Principal Investigator, Xiuhua Sun, Chief physician, Dalian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-BV-MCL
Record Dates: First submitted 2024-03-09; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: Linperlisib; Venetoclax; Obinutuzumab
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort 1 (Experimental): Patients with relapsed refractory lymphoblastic mantle cell lymphoma who have not previously received treatment with PI3K inhibitors and BCL-2 inhibitors
  Interventions: Drug: Linperlisib in combination with Obinutuzumab and Venetoclax

INTERVENTIONS:
Drug: Linperlisib in combination with Obinutuzumab and Venetoclax — Combined induction period: Linprixate: 80 mg, oral (pre - and post meal), once a day; Otuzumab: 1000 mg/dose, intravenous infusion, administered on the first day (1st cycle is 1, 8, 15 days); (Up to 6 cycles, administration cycle can be adjusted according to clinical treatment conditions); Vineclavone: increase from 40mg, 100mg, and 200mg to 400mg within 4 weeks, followed by a treatment cycle of 400mg orally once a day; (Starting from the third cycle), one cycle every 28 days, for a total of 6 cycles。 Maintenance treatment period: Linprixate: 80 mg, oral (both before and after meals), once a day; Vinecala: 400 mg, oral, once daily; Cycle every 28 days.
  Other Names: Treatment group

SUMMARY:
This is a single arm, open label, national multicenter clinical study included patients with relapsed and refractory blastoid variant of mantle cell lymphoma (R/R BV-MCL), aiming to evaluate the efficacy of a chemotherapy free triple therapy of PI3K inhibitor (Linperlisib) combined with anti-CD20 monoclonal antibody (Obinutuzumab) and BCL-2 inhibitor (Venetoclax) in R/R BV-MCL patients.

DETAILED DESCRIPTION:
This is a single arm, open label, national multicenter clinical study that included 10 cases of relapsed and refractory blastoid variant of mantle cell lymphoma (R/R BV-MCL). The aim was to evaluate the efficacy of a chemotherapy free triple therapy consisting of PI3K inhibitor (Linperlisib) combined with anti-CD20 monoclonal antibody (Obinutuzumab) and BCL-2 inhibitor (Venetoclax) in patients with R/R BV-MCL. It is divided into a combined induction period and a maintenance treatment period. All enrolled patients receive the following combined treatment: combined induction period: Linperlisib: 80 mg, orally (pre - and post meal), once a day; Obinutuzumab: 1000 mg/dose, intravenous infusion, administered on the first day (1st cycle is 1, 8, 15 days); (Up to 6 cycles, administration cycle can be adjusted according to clinical treatment conditions); Venetoclax: increase from 40mg, 100mg, and 200mg to 400mg within 4 weeks, followed by a treatment cycle of 400mg orally once a day; (Starting from the third cycle). Every 28 days, there are a total of 6 cycles. Maintenance treatment period: Linperlisib: 80 mg, oral (both before and after meals), once a day; Venetoclax: 400 mg, oral, once daily. Cycle every 28 days. After 6 cycles of combined treatment, the efficacy is evaluated according to the Lugano2014 standard. If complete remission (CR) or partial remission (PR) is achieved, maintenance treatment with a combination of 80 mg of linprixate and 400 mg of vinclair is administered every 28 days until disease progression, intolerable toxicity, or other reasons lead to discontinuation. If it is stable disease (SD) and progressive disease (PD), patients will be excluded from the group. The main research endpoint is Objective Response Rate (ORR). Secondary study endpoints include progression free survival (PFS); Overall survival (OS), duration of response (DOR), and safety: incidence and severity of adverse events (AE) and severe adverse events (SAE). Safety: incidence and severity of adverse events (AE) and severe adverse events (SAE).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Mother cell type mantle cell lymphoma (BV-MCL) confirmed by histopathological and immunophenotypic analysis;
* The Eastern Oncology Collaborative Group (ECOG) scored 0-2 on physical fitness status;
* Expected lifespan ≥ 3 months
* There is at least one measurable lesion: the longest diameter (LDi) of lymph node lesions is ≥ 1.5 cm, or the LDi of extralymph node lesions is ≥ 1 cm, or splenomegaly, or bone marrow involvement with or without malignant lymphocytosis;
* Have not received treatment with PI3K inhibitors and BCL-2 inhibitors in the past; Having sufficient bone marrow and organ functions;
* Having sufficient bone marrow and organ functions;
* All screening period laboratory tests must be conducted according to the requirements of the plan, and must be conducted within 7 days before enrollment. The values of laboratory tests conducted for screening must meet the following criteria:

Blood routine examination (no blood transfusion, no use of granulocyte colony-stimulating factor (G-CSF), no medication correction within 14 days prior to screening):

1. Hemoglobin (Hb) ≥ 80 g/L;
2. Neutrophils (ANC) ≥ 1.0 × 109/L;
3. Platelet count (PLT) ≥ 75 × 109/L;

Biochemical examination:

1. TBIL<1.5 × Upper limit of normal range (ULN);
2. Glutamate alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN;
3. Serum creatinine (Cr) ≤ 1.25 × ULN or endogenous creatinine clearance rate ≥ 60 mL/min (Cockcroft Gault formula);

Coagulation function (unless the subject is receiving anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant therapy at the time of screening):

1. International normalized ratio (INR) ≤ 1.5 × ULN;
2. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;

   * Those who have not participated in clinical trials of other drugs within the 4 weeks prior to enrollment;
   * Women with a possibility of pregnancy must undergo a serum pregnancy test within 7 days before the first medication, and the result is negative. They are willing to Intended to use efficient methods of contraception during the trial period and within 1 year after the last administration of the investigational drug. For male subjects whose partners are women of childbearing age, they should undergo surgical sterilization or agree to use high-efficiency contraception methods during the trial period and 1 year after the last administration of the trial drug;
   * The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Patients who have received any targeted PI3K or BCL treatment before enrollment;
* History of other primary invasive malignant tumors that have not been relieved or have not been relieved for more than 3 years;
* Those with involvement of the central nervous system (meninges or brain parenchyma);
* Individuals who are known to have allergies to any medication in the study;
* Participated in clinical trials of other drugs within 4 weeks prior to the start of the study;
* Pregnant or lactating women;
* Individuals with active infections, excluding fever related to tumor B symptoms;
* Concomitant diseases and medical history:

  1. There are multiple factors that affect oral medication, such as inability to swallow, chronic diarrhea, and intestinal obstruction
  2. Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
  3. Subjects with any severe and/or uncontrolled diseases, including:

     1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
     2. Suffering from ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia [including QTc ≥ 450ms (male), QTc ≥ 470ms (female)], and ≥ grade 2 congestive heart failure [NYHA classification];
     3. Active interstitial pneumonia or other chronic lung diseases leading to severe impairment of lung function, defined as FEV1 and DLCOc<60% of normal predicted values;
     4. Liver abnormalities;
     5. Decompensated cirrhosis (Child Pugh liver function rating of B or C)
     6. Known clinically significant history of liver disease. Including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e. HBV DNA positivity (>2500 copies/mL or>500 IU/mL, and above the upper limit of normal values); Known hepatitis C virus infection (HCV) and HCV RNA positivity (>1×103copies/mL). Note: hepatitis B HBsAg positive subjects who meet the inclusion conditions, whether their HBV DNA is measurable or not, need to continue antiviral treatment (nucleoside analogues are recommended) and regularly monitor HBV DNA; For subjects with positive HBcAb but negative HBsAg in hepatitis B, HBV DNA should be monitored regularly and preventive antiviral treatment should be recommended; Hepatitis C patients need to regularly monitor HCV RNA.
     7. Renal failure requiring hemodialysis or peritoneal dialysis;
     8. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
     9. Poor control of diabetes (FBG>10 mmol/L);
     10. Urine routine indicates urine protein ≥++, and it is confirmed that the 24-hour urine protein quantification is greater than 1.0 g;
* Have a history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* According to the researcher's judgment, there are accompanying diseases that seriously endanger patient safety or affect patient completion of the study. Unable to understand the nature of the research or disagrees to sign an informed consent form;
* The researcher evaluates other situations that are not suitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to the RECIST 1.1 | At the end of Cycle 6 (each cycle is 28 days)
  The ORR rate of patients with Linperlisib in combination with Obinutuzumab and Venetoclax for relapsed and refractory blastoid variant of mantle cell lymphom

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of enrollment until the date of first documented progression and loss of follow-up or date of death from any cause, whichever came first, assessed up to 24 months
  The time from the start of clinical trials to the occurrence (in any aspect) of tumor progression or death due to any reason
Overall survival (OS) | From date of enrollment until the date of first date of death from any cause, expected evaluation period of up to 48 months
  The time from the start of tumor treatment to (for any reason) death.
Duration of Overall Response (DOR) | From date of the time from the first assessment of the tumor as CR or PR to the first assessment as PD (Progressive Disease) or death from any cause,assessed up to 24 months
  The time from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD).
Adverse event (AE) | Record any adverse events starting from the first medication use until the end of the safety follow-up period. The evaluation period shall not exceed 24 months.
  Refers to adverse medical events that occur in the clinical trial process of the subject

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Sun, Doctor, Study Director — Dalian Medical University
Locations (1):
- The Second Hospital Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No